CLINICAL TRIAL: NCT00298532
Title: The Ontario Prehospital Advanced Life Support (OPALS) Study for Critically Ill and Injured Pediatric Patients
Brief Title: OPALS Pediatric Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Ian G. Stiell, Principal Investigator, Ottawa Hospital Research Institute
Allocation: Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: MOP 64269
Record Dates: First submitted 2006-03-01; First posted 2006-03-02 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2010-10

CONDITIONS: Seizure
Keywords: Pediatrics; Seizure; Trauma; Respiratory; Cardiac; Arrest
MeSH Terms: conditions — Seizures; Wounds and Injuries; Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- standard therapy (No Intervention): The use of a before-after controlled study design and 36-month time periods will mirror the approach of our Adult OPALS Study. The Control (before) Period represents the 36 months immediately prior to the introduction of ALS programs at each study community. The Intervention (after) Period is comprised of the 36 months immediately after each community has met all standards for a full ALS program, as defined below. Data will be pooled across communities but the start date for the periods will vary for each community as each will require different amounts of time to prepare their ALS program. A 6- to 36-month "Run-in" period will separate the Control and Intervention Periods and will allow for training and implementation of the ALS program. Data from the Run-in period will not be considered in the primary analysis. The study periods may be summarized as follows: a) Control (Before) Period b) Run-in Period c) Intervention (After) Period.
  Interventions: Procedure: Advanced Life Support

INTERVENTIONS:
Procedure: Advanced Life Support

SUMMARY:
The OPALS Pediatric Study will examine the incremental impact of introducing a prehospital full advanced life support in pediatric patients.

DETAILED DESCRIPTION:
Background: Pediatric patients constitute a significant proportion of all ambulance transports by emergency medical services (EMS) with the most common conditions being trauma, respiratory distress, and seizures. Cardiopulmonary arrest is a less common condition but has a mortality rate in children in excess of 98%. Very little evidence is available regarding the effectiveness of prehospital interventions for children. Canadian communities require guidance as to whether their local EMS services should implement full advanced life support (ALS) measures for pediatric patients. This proposal builds upon the Adult OPALS Study, the largest controlled out-of-hospital study ever conducted worldwide, which is evaluating the impact of ALS programs in multiple Ontario cities on 35,000 adult patients.

Objectives: The goal of the Pediatric OPALS Study is to evaluate the benefit of introducing a prehospital program of full ALS measures (intubation and intravenous drug therapy) on the outcomes of critically ill and injured pediatric patients. Specific objectives are to determine the impact of this ALS program on mortality, other clinical outcomes, morbidity (quality of life), EMS response intervals, and cost-effectiveness for these critical conditions: a) Respiratory distress and obstruction, b) Seizure, c) Major trauma, and d) Cardio-pulmonary arrest. We hypothesize, for each of the four patient populations separately, that in the Intervention period: i) Mortality will be reduced (primary hypothesis); ii) Other Clinical Measures will be improved for other clinical outcomes, ED interventions, admission rates, and lengths of stay; iii) Quality of Life of survivors will be improved for both generic and disease-specific measures; iv) Response Time Intervals will not be increased; and, v) Economic Evaluation will reveal that the costs and effects are distributed more favourably.

Methods: The Pediatric OPALS Study will incorporate a before-after design with the unit of study being all eligible patients seen during each of two distinct 36-month periods in 17 Ontario cities. During the baseline Control (Before) Period (1992-1998), the study cities provided BLS-D level of care with first-responder firefighters and Primary Care Paramedics. During the Intervention (After) Period (1998-2002), the study cities provided a full pre-hospital ALS program. The study population is all patients under the age of 16 years who were treated out-of-hospital for any of these four conditions: a) Respiratory Distress or Obstruction, defined as patients with a chief complaint of shortness of breath, respiratory arrest, or airway obstruction; b) Seizure, defined as patients having suffered a generalized convulsion; c) Major Trauma, defined as patients with injuries caused by any mechanism and associated with an Injury Severity Score (ISS) more than 12; d) Cardiopulmonary Arrest, defined as patients with absence of a detectable pulse, unresponsiveness, and apnea. The study intervention was implemented during the "Run-in" period, immediately prior to the Intervention period, and entails a program of pre-hospital ALS care provided by EMS: a) Endotracheal Intubation, b) Intravenous therapy, and c) Administration of intravenous drugs. Study cities had to meet four strict performance criteria. Data will be obtained by electronic or hard copy means from the following sources: Ambulance Call Reports, Fire Medical Reports, Base Hospital Reviews, Ambulance Response Information System, Hospital Records, Ontario Trauma Registry, and Follow-up Interviews. The primary outcome measure will be mortality. Secondary outcomes include a) Other Clinical Measures (Other Survival, Need for Interventions in the ED, Admission, Lengths of Stay), b) Generic Quality of Life (HUI3), c) Disease-specific Quality of Life (CPC, FIM), d) Response Time Intervals, and g) Direct Costs. The primary data analysis will test the hypothesis that mortality discharge will be improved when comparing the after period to the before period by chi-square analysis techniques. Stepwise logistic regression analysis will be performed to control for the possible confounding effects of various indicators and to assess the effect of the study period on survival. The study will involve a total of 18,000 pediatric patients over 72 months.

Importance: This proposed study has a unique opportunity to evaluate the effectiveness of ALS interventions on the outcomes of critically ill and injured patients. Never again may there be such an opportunity to conduct a controlled evaluation of the impact of an ALS program in such a large population. The results of this study will be very important to health care planners in Canada and throughout the world.

ELIGIBILITY:
Inclusion Criteria:

* Patients less than 16 years of age transported to the Emergency Department with either seizure, acute trauma, respiratory distress or cardiac arrest.

Exclusion Criteria:

* Patients over 16 years of age or older.

Ages: 1 Day to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9000
Dates: Start 1992-07; Primary Completion 2007-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Survival to discharge Quality of life Response time intervals Performance of ALS intervals Emergency department interventions Admission rates Length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Ian Stiell, MD, Principal Investigator — OHRI
Locations (10):
- Canada (10):
  - Cambrige Base Hospital, Cambridge, Ontario
  - Sudbury Base Hospital, Greater Sudbury, Ontario
  - Kingston Base Hospital, Kingston, Ontario
  - London Base Hospital, London, Ontario
  - Halton Base Hospital, Mississauga, Ontario
  - Niagara Falls Base Hospital, Niagara Falls, Ontario
  - Ottawa Base Hospital, Ottawa, Ontario
  - Peterborough Base Hospital, Peterborough, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - Hotel Dieu Grace Hospital, Windsor, Ontario